CLINICAL TRIAL: NCT02337387
Title: A Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of 2 Formulations of Blosozumab in Postmenopausal Women
Brief Title: A Study of 2 Different Formulations of Blosozumab (LY2541546) in Post Menopausal Women
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol stopping criteria (safety) were met.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 15728; I2M-MC-GSDT (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — blosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Blosozumab Formulation A (Experimental): Part A. Blosozumab administered as 2 subcutaneous (SC) injections in week 1 followed by once weekly (QW) injections SC in weeks 2 to 6, followed by six week follow-up period.
  Interventions: Biological: Blosozumab
- Blosozumab Formulation B (Experimental): Part A. Blosozumab administered as 2 SC injections in week 1 followed by QW injections SC in weeks 2 to 6, followed by six week follow-up period.
  Interventions: Biological: Blosozumab
- Placebo (Placebo Comparator): Part A. Placebo administered as 2 SC injections in week 1 followed by QW injections SC in weeks 2 to 6, followed by six week follow-up period.
  Interventions: Other: Placebo
- Blosozumab (Part B) (Experimental): Part B. Blosozumab formulation determined by Part A administered as 2 SC injections in week 1 followed by QW injections SC in weeks 2 to 6, followed by six week follow-up period.
  Interventions: Biological: Blosozumab

INTERVENTIONS:
Biological: Blosozumab — Administered SC
  Other Names: LY2541546
  Arms: Blosozumab (Part B); Blosozumab Formulation A; Blosozumab Formulation B
Other: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the tolerability of two different formulations of blosozumab in women who have reached menopause.

This study will last approximately 12 weeks for each participant, not including screening. Screening is required within 28 days prior to starting the study.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Overtly healthy postmenopausal (PMP) females
* Part B: PMP women who are currently taking oral bisphosphonates for prevention or treatment of osteoporosis
* Have a body mass index (BMI) at screening of 19.0 to 35.0 kilogram per square meter (kg/m^2)

Exclusion Criteria:

* Have known allergies to blosozumab, its constituents, or related compounds
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* History of breast carcinoma
* Fracture of a long bone within 1 year of screening
* Have used teriparatide within 3 years prior to screening

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Covance, Daytona Beach, Florida
  - Covance Clinical Research Inc, Evansville, Indiana
  - Covance, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was designed to have two parts. During Part A, one participant in each blosozumab treatment arm developed non-serious AEs, which met criteria for stopping the study. One participant was discontinued from the trial due to this AE. All other participants were discontinued due to trial termination. Part B was not conducted.
Groups:
- Blosozumab Formulation A: Part A - Blosozumab Formulation A administered as a 180 milligram (mg) loading dose subcutaneously (SC) in Week 1 followed by 90 mg SC once weekly (QW) for 5 weeks. Participants were followed for 7 weeks after the last dose.
- Blosozumab Formulation B: Part A - Blosozumab Formulation B administered as a 180 mg loading dose SC in Week 1 followed by 90 mg SC QW for 5 weeks. Participants were followed for 7 weeks after the last dose.
- Placebo Formulation A: Part A - Placebo matching Blosozumab Formulation A administered as a loading dose SC in Week 1 followed by a SC injection QW for 5 weeks. Participants were followed for 7 weeks after the last dose.
- Placebo Formulation B: Part A - Placebo matching Blosozumab Formulation B administered as a loading dose SC in Week 1 followed by a SC injection QW for 5 weeks. Participants were followed for 7 weeks after the last dose.
Period: Overall Study
Arm/Group | Blosozumab Formulation A | Blosozumab Formulation B | Placebo Formulation A | Placebo Formulation B
Started | 14 | 8 | 3 | 3
Received at Least 1 Dose of Study Drug | 14 | 8 | 3 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 14 | 8 | 3 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Sponsor Decision to Terminate Study | 14 | 7 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Blosozumab Formulation A: Blosozumab Formulation A administered as a 180 mg loading dose SC in Week 1 followed by 90 mg SC QW for 5 weeks. Participants were followed for 7 weeks after the last dose.
- Blosozumab Formulation B: Blosozumab Formulation B administered as a 180 mg loading dose SC in Week 1 followed by 90 mg SC QW for 5 weeks. Participants were followed for 7 weeks after the last dose.
- Placebo Formulation A: Placebo matching Blosozumab Formulation A administered as a loading dose SC in Week 1 followed by a SC injection QW for 5 weeks. Participants were followed for 7 weeks after the last dose.
- Placebo Formulation B: Placebo matching Blosozumab Formulation B administered as a loading dose SC in Week 1 followed by a SC injection QW for 5 weeks. Participants were followed for 7 weeks after the last dose.
- Total: Total of all reporting groups
Arm/Group | Blosozumab Formulation A | Blosozumab Formulation B | Placebo Formulation A | Placebo Formulation B | Total
Number analyzed (Participants) | 14 | 8 | 3 | 3 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (4.3) | 58.1 (5.0) | 56.3 (4.6) | 56.0 (9.8) | 58.3 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 3 | 3 | 28
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 2 | 0 | 10
  Not Hispanic or Latino | 8 | 6 | 1 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 3
  White | 12 | 7 | 2 | 1 | 22
  More than one race | 0 | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 8 | 3 | 3 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other nonserious adverse events (AEs) and all SAEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through Day 85
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Blosozumab Formulation A | Blosozumab Formulation B | Placebo Formulation A | Placebo Formulation B
Number analyzed (Participants) | 14 | 8 | 3 | 3
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Blosozumab Formulations A and B
Time Frame: Day 1: Predose, 24 Hours (H), 72 H, 120 H, 168 H Post Loading Dose
Population: All participants who received the loading dose of blosozumab and had evaluable Cmax values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per milliliter (pmol/mL)
Arm/Group | Blosozumab Formulation A | Blosozumab Formulation B
Number analyzed (Participants) | 14 | 8
picomoles per milliliter (pmol/mL) | 63.4 (82) | 51.0 (108)

3. Secondary Outcome: Pharmacokinetics: Time to Maximum Concentration (Tmax) of Blosozumab Formulations A and B
Time Frame: Day 1: Predose, 24 Hours (H), 72 H, 120 H, 168 H Post Loading Dose
Population: All participants who received the loading dose of blosozumab and had evaluable Tmax values.
Measure: Median (Full Range); unit: hours
Arm/Group | Blosozumab Formulation A | Blosozumab Formulation B
Number analyzed (Participants) | 14 | 8
hours | 120 [72 to 168] | 120 [72 to 168]

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve During 1 Dosing Interval (AUC[0-tau]) of Blosozumab Formulations A and B
Time Frame: Day 1: Predose, 24 Hours (H), 72 H, 120 H, 168 H Post Loading Dose
Population: All participants who received the loading dose of blosozumab and had evaluable AUC(0-tau) values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*hours per mL
Arm/Group | Blosozumab Formulation A | Blosozumab Formulation B
Number analyzed (Participants) | 14 | 8
pmol*hours per mL | 7880 (83) | 6400 (110)

ADVERSE EVENTS:
Time Frame: Baseline through Day 85
Description: Includes SAEs and all other non-serious AEs that met the frequency threshold regardless of causality. Non-serious AEs met criteria for stopping the study.
Arm/Group | Blosozumab Formulation A | Blosozumab Formulation B | Placebo Formulation A | Placebo Formulation B
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 11/14 | 5/8 | 2/3 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blosozumab Formulation A (N=14) | Blosozumab Formulation B (N=8) | Placebo Formulation A (N=3) | Placebo Formulation B (N=3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 6 (11) | 3 (5) | 1 (3) | 0 (0)
Injection site discolouration (General disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 11 (35) | 5 (11) | 2 (4) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 5 (9) | 1 (2) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 6 (12) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Protocol stopping criteria (safety) were met. Non-serious AEs met criteria for stopping the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days